CLINICAL TRIAL: NCT03083379
Title: A Pilot Evaluation Comparing Regional Distribution of Ventilation During Lung Expansion Therapy in Healthy Adult Human Subjects
Brief Title: Pilot Evaluation Comparing Regional Distribution of Ventilation During Lung Expansion Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Draeger Medical, Inc (Industry)
Responsible Party: Principal Investigator, Daniel D Rowley, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19661
Record Dates: First submitted 2017-03-06; First posted 2017-03-20 (Actual); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Ventilation; Breathing; Atelectasis
Keywords: Incentive spirometry; EzPAP; Electrical impedance tomography
MeSH Terms: conditions — Respiratory Aspiration; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Volumetric Incentive Spirometry (Active Comparator): Incentive Spirometry
  Interventions: Device: Volumetric Incentive Spirometry
- EzPAP® POSITIVE AIRWAY PRESSURE (Experimental): EzPAP
  Interventions: Device: EzPAP® POSITIVE AIRWAY PRESSURE

INTERVENTIONS:
Device: Volumetric Incentive Spirometry — A study investigator will provide instruction on Incentive Spirometry procedure performance before supervised therapy and monitoring begins.
  * Five minutes of eupneic ventilation EIT monitoring will occur before I.S. therapy commences.
  * Study participants will be asked to take 10 deep breaths through the incentive spirometer's mouthpiece, followed by a 60 second pause.
  * The 10-breath cycle will be repeated three times with respiratory therapist coaching.
  * Five minutes of eupneic ventilation EIT monitoring will occur following the last I.S. lung expansion therapy breath cycle.
  * Incentive Spirometry therapy and monitoring session will last about 15 minutes
  Other Names: I.S.
  Arms: Volumetric Incentive Spirometry
Device: EzPAP® POSITIVE AIRWAY PRESSURE — * A study investigator will provide instruction on EzPAP® procedure performance before supervised therapy and monitoring begins. A second study investigator will perform EIT device set-up and monitoring only.
  * Five minutes of eupneic ventilation EIT monitoring will occur before EzPAP® therapy commences.
  * Study participants will be asked to breathe normally through the EzPAP® device's mouthpiece for 10 breaths, followed by a 60 second pause.
  * The 10-breath cycle will be repeated three times with respiratory therapist coaching.
  * Five minutes of eupneic ventilation EIT monitoring will occur following the last EzPAP® lung expansion therapy breath cycle.
  * EzPAP® therapy and monitoring sessions will last about 15 minutes
  Other Names: EzPAP®
  Arms: EzPAP® POSITIVE AIRWAY PRESSURE

SUMMARY:
The primary purpose of this study is to determine if there is a significant difference in regional distribution of ventilation when comparing eupneic tidal ventilation with Incentive Spirometry (I.S.) and EzPAP® lung expansion therapy in healthy adult human subjects. Electrical impedance tomography (EIT) will be used to measure regional distribution of ventilation during resting tidal ventilation and during lung expansion therapy.

DETAILED DESCRIPTION:
Investigators will use a convenience sampling scheme to identify potential study participants. Documentation of informed consent will be recorded. Electrical Impedance Tomography (Pulmovista 500; Draeger, Lubeck, Germany), which provides non-invasive and radiation free monitoring, will be used to monitor and measure regional distribution of ventilation during I.S and EzPAP® lung expansion therapy.

Recruitment email will be will be sent to University of Virginia Medical Center employees who represent the target study population. A university of Virginia email distribution list will be used to mass email respiratory therapy and nursing staff working in adult ICU and surgical acute care patient wards. Word of mouth will also be used to heighten awareness about this study.

A computer generated random numbers generator will be used to randomly assign study subjects into an I.S. or EzPAP® lung expansion therapy group after documentation of informed consent has been recorded. Randomization masking/blinding will not occur in this study. The lung expansion therapy medical device designs and their respective operational differences are impossible to conceal.

Procedure set-up and device calibration will occur according to Draeger provided PulmoVista 500 (Draeger; Lubeck, Germany) EIT training and operation manual:

* Study participant preparation

  * Investigator will select an electrode belt and respective patient cable sizes after measuring participant's chest circumference with paper measurement tape placed across the midclavicular line at intercostal space 4 -5. Electrode belt size will be selected according to a chest circumference measurement that aligns best to the manufacturer's recommended belt size identified in a belt selection table.
  * A patient cable of the same electrode belt size will be selected and connected to the electrode belt before connection to study participants. Investigator will align and snap connect the patient cable snaps over the electrode belt studs by aligning respective snaps and studs in ascending numerical order from 1 to 16.
  * A light spray of warm tap water will be applied to the electrode surface on the electrode belt before it is applied to study participants to optimize conductivity between the skin and electrodes.
* Attaching electrode belt and reference electrode to study participant while they are positioned at 45-degrees sitting in a reclining chair.

  * The electrode belt/cable combination will be attached around the thorax of each study participant at the level of the 4th - 5th intercostal space, unless mammary tissue prevents this site of application. An alternative application site will be located immediately below the mammary tissue if necessary. Left to right belt orientation will be maintained with color coded patient cable ports signifying left and right side.
  * An investigator will snap the electrode belt closed after verifying proper belt position. The belt's black electrodes should have close contact with the study participant's skin at this point.
  * An adhesive ECG electrode will be place on the study participant's right upper abdominal quadrant and then the patient cable reference electrode snap will be attached to the ECG electrode.
  * The patient cable will then be connected to the EIT monitoring device (PulmoVista 500, Lubeck, Germany) via a color coded trunk cable orientation that aligns with the patient cable left and right orientation.
* EIT device calibration and signal check

  * Investigator will initiate a PulmonVista 500 EIT monitoring device calibration each day prior to performing new study participant EELI measurements.
  * A skin-electrode signal check will be performed to ensure that a minimum of 15 of 16 electrodes have sufficient contact with the participant's skin surface and signal quality is stable.
* Monitoring sessions and Lung Expansion Therapy procedure

  * Monitoring will be initiated after researcher performs PulmoVista 500 EIT device (Draeger; Lubeck, Germany) setup and calibration.
  * Approximate monitoring/measurement duration is 15-minutes.

INCENTIVE SPIROMETRY GROUP

- A study investigator will instruct the study participant to strive for an inspiratory capacity volume target as determined by the I.S. device's predicted volume nomogram table.

Incentive Spirometry procedure A study investigator will provide instruction on Incentive Spirometry procedure performance before supervised therapy and monitoring begins.

* Five minutes of eupneic ventilation EIT monitoring will occur before I.S. therapy commences.
* Study participants will be asked to take 10 deep breaths through the incentive spirometer's mouthpiece, followed by a 60 second pause.
* The 10-breath cycle will be repeated three times with respiratory therapist coaching.
* Five minutes of eupneic ventilation EIT monitoring will occur following the last I.S. lung expansion therapy breath cycle.
* Incentive Spirometry therapy and monitoring session will last about 15 minutes.

EzPAP® POSITIVE AIRWAY PRESSURE GROUP

* A study investigator will provide instruction on EzPAP® procedure performance before supervised therapy and monitoring begins. A second study investigator will perform EIT device set-up and monitoring only.
* Five minutes of eupneic ventilation EIT monitoring will occur before EzPAP® therapy commences.
* Study participants will be asked to breathe normally through the EzPAP® device's mouthpiece for 10 breaths, followed by a 60 second pause.
* The 10-breath cycle will be repeated three times with respiratory therapist coaching.
* Five minutes of eupneic ventilation EIT monitoring will occur following the last EzPAP® lung expansion therapy breath cycle.
* EzPAP® therapy and monitoring sessions will last about 15 minutes.

REGIONAL DISTRIBUTION OF VENTILATION MONITORING:

* PulmoVista monitoring and lung expansion therapy will occur only one time as described above.
* Global and regional distribution of ventilation data will be displayed on the PulmoVista 500 device's main monitoring screen during lung expansion therapy, but study investigator staff administering therapy and study participants will be blinded from information displayed on the screen's monitor during therapy session in an effort to reduce performance bias.

  * Once lung expansion therapy session has ended, the investigator will detach trunk cables from electrode cables, detach reference electrode snap from adhesive ECG electrode, unclamp the electrode belt, and then remove belt from the study participant. Subject participation in this study is considered complete at this time.
  * Inspection of electrode belt contact area will be performed to assess for evidence of skin irritation or bruising. Study participant will be notified by study investigator at the time of skin assessment if significant skin irritation or bruising is present. Finding will be recorded by study investigator.
* Electrode belt, patient cable, and PulmoVista 500 EIT device (Draeger; Lubeck, Germany) will be removed study participant's room and returned to a storage location outside of patient care areas.
* Following each EIT to subject interface disconnect, an alcohol, aldehyde, or quaternary ammonium based compound will be soaked on a wipe cloth to disinfect the surfaces of the patient cable, electrode belt, trunk cable, and EIT unit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy- not receiving in-patient medical care
* Documentation of written informed consent

Exclusion Criteria:

* Less than 18 or greater than 79 years of age
* Body mass index > 50
* Excessive chest hair
* Inability to obtain written informed consent
* Inability to follow verbal instructions
* Pregnancy: self reported
* Uncontrolled body movements
* Inability to place EIT electrodes and belt in direct contact with skin where they are projected to come into contact
* Active implants (i.e., cardiac pacemaker, implantable cardioverter-defibrillator [ICD]), or when device compatibility is in doubt.)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Rowley, MSc RRT-ACCS, Principal Investigator — Pulmonary Diagnostics & Respiratory Therapy Servies, University of Virginia Medical Center
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Volumetric Incentive Spirometry: Incentive Spirometry
  Volumetric Incentive Spirometry: A study investigator will provide instruction on Incentive Spirometry procedure performance before supervised therapy and monitoring begins.
  * Five minutes of eupneic ventilation EIT monitoring will occur before I.S. therapy commences.
  * Study participants will be asked to take 10 deep breaths through the incentive spirometer's mouthpiece, followed by a 60 second pause.
  * The 10-breath cycle will be repeated three times with respiratory therapist coaching.
  * Five minutes of eupneic ventilation EIT monitoring will occur following the last I.S. lung expansion therapy breath cycle.
  * Incentive Spirometry therapy and monitoring session will last about 15 minutes
- EzPAP® POSITIVE AIRWAY PRESSURE: EzPAP
  EzPAP® POSITIVE AIRWAY PRESSURE: - A study investigator will provide instruction on EzPAP® procedure performance before supervised therapy and monitoring begins. A second study investigator will perform EIT device set-up and monitoring only.
  * Five minutes of eupneic ventilation EIT monitoring will occur before EzPAP® therapy commences.
  * Study participants will be asked to breathe normally through the EzPAP® device's mouthpiece for 10 breaths, followed by a 60 second pause.
  * The 10-breath cycle will be repeated three times with respiratory therapist coaching.
  * Five minutes of eupneic ventilation EIT monitoring will occur following the last EzPAP® lung expansion therapy breath cycle.
  * EzPAP® therapy and monitoring sessions will last about 15 minutes
Period: Overall Study
Arm/Group | Volumetric Incentive Spirometry | EzPAP® POSITIVE AIRWAY PRESSURE
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Volumetric Incentive Spirometry | EzPAP® POSITIVE AIRWAY PRESSURE | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [28 to 55] | 31 [27 to 45] | 35 [28 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Change in dorsal regional distribution of ventilation [Median (Inter-Quartile Range); unit: Percent] | 2.9 [-2.6 to 9.4] | 2.8 [-0.3 to 4.6] | 2.8 [-0.78 to 6.4]

OUTCOME MEASURES:

1. Primary Outcome: Regional Distribution of Ventilation
Description: EIT will be used to measure change in regional distribution of ventilation during lung expansion therapy.
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: percentage of dorsal redistribution
Arm/Group | Volumetric Incentive Spirometry | EzPAP® POSITIVE AIRWAY PRESSURE
Number analyzed (Participants) | 15 | 15
percentage of dorsal redistribution | -4.9 [-15.9 to 6.0] | -5.6 [-14.0 to 2.7]
Statistical Analysis 1: Comparison: Volumetric Incentive Spirometry vs EzPAP® POSITIVE AIRWAY PRESSURE; Test type: Equivalence — Equivalency is defined as no statistically significant difference in dorsal region redistribution of ventilation following breath cycle 1, 2, and 3 lung expansion therapy sequences; p = .90, Mann-Whitney U test

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Volumetric Incentive Spirometry | EzPAP® POSITIVE AIRWAY PRESSURE
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
This was a pilot study with a small enrollment sample. Study is underpowered to detect statistical significance if one exists between the primary group compared outcome measurement; Dorsal percent change in redistribution of ventilation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03083379/Prot_SAP_000.pdf